CLINICAL TRIAL: NCT01120886
Title: Post-mortem Genetic Testing for Cardiac Ion Channelopathy in Unexplained Still Births
Brief Title: Post-mortem Genetic Testing
Status: Completed | Type: Observational
Sponsor: Thayyil, Sudhin (Individual)
Responsible Party: Principal Investigator, Sudhin Thayyil, Consultant Neonatologist, Thayyil, Sudhin
Other Study IDs: 48699
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Cardiac Ion Channelopathy
Keywords: Ion channelopathy,; Still birth; Sudden death
MeSH Terms: conditions — Stillbirth; Death, Sudden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin and muscle
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective observational study to examine the incidence of cardiac ion channelopathies in unexplained still births.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained still births,
* No cause of death after detailed autopsy

Exclusion Criteria:

* Lack of parental consent

Ages: 24 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Unexplained still births
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Incidence of cardiac ion channelopathy mutation | 6 months

SECONDARY OUTCOMES:
Incidence of cardiac ion channelopathy in 1st degree relatives of index case | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - Southampton University Hospital, Southampton

REFERENCES:
- [Derived] Munroe PB, Addison S, Abrams DJ, Sebire NJ, Cartwright J, Donaldson I, Cohen MM, Mein C, Tinker A, Harmer SC, Aziz Q, Terry A, Struebig M, Warren HR, Vadgama B, Fowler DJ, Peebles D, Taylor AM, Lally PJ, Thayyil S. Postmortem Genetic Testing for Cardiac Ion Channelopathies in Stillbirths. Circ Genom Precis Med. 2018 Jan;11(1):e001817. doi: 10.1161/CIRCGEN.117.001817. Epub 2018 Jan 11. PMID 29874177
- See also: Institute for Women's Health — http://www.instituteforwomenshealth.ucl.ac.uk/academic_research/neonatology/pm-mri